CLINICAL TRIAL: NCT02194387
Title: Pilot Tests to Optimize the Delivery of Energy Balance Interventions
Brief Title: Energy Balance Interventions in Increasing Physical Activity in Breast Cancer Gene Positive Patients, Lynch Syndrome-Positive Patients, CLL Survivors or High-Risk Family Members
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-0230; NCI-2015-00095 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0230 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Body Mass Index 25 or Greater; BRCA1 Gene Mutation; BRCA2 Gene Mutation; Breast Carcinoma; Cancer Survivor; Chronic Lymphocytic Leukemia; Fatigue; Health Status Unknown; Lynch Syndrome; Ovarian Carcinoma; Overweight
MeSH Terms: conditions — Breast Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Fatigue; Colorectal Neoplasms, Hereditary Nonpolyposis; Ovarian Neoplasms; Overweight | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (energy balance interventions) (Experimental): TELEPHONE COACHING VS EMAIL COACHING: Participants receive telephone coaching once per week for 16 weeks or 1 email per week for 16 weeks (with follow-up responses if the participant responds) from a coach trained in motivational interviewing.
  TEXT MESSAGES: Participants receive daily text messages promoting adherence to diet and exercise recommendations daily 1-3 times per day or no text messages.
  SOCIAL NETWORKING: Participants are invited to an online forum for study participants available for 16 weeks or do not receive an invitation for social networking.
  SELF-MONITORING: Participants are asked to record their dietary intake 4-7 days per week or 1 day per week on a website or smartphone app.
  Interventions: Dietary Supplement: Dietary Intervention; Other: Internet-Based Intervention; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Record dietary intake 4-7 days per week
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Dietary Supplement: Dietary Intervention — Record dietary intake 1 day per week
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Other: Internet-Based Intervention — Receive email coaching
Other: Internet-Based Intervention — Participate in social networking
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive telephone coaching
Behavioral: Telephone-Based Intervention — Receive text messages

SUMMARY:
This pilot clinical trial studies different types of energy balance interventions to see how well they work in increasing the physical activity levels of breast cancer gene-positive patients, Lynch syndrome-positive patients, chronic lymphocytic leukemia (CLL) survivors or family members of cancer survivors who are at high risk for cancer. Increasing exercise and eating healthy foods may help reduce the risk of cancer. Studying how well different types of interventions work in motivating cancer survivors or high-risk family members to increase exercise and healthy food choices may help doctors plan the most effective motivational program for cancer prevention.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the feasibility of using the multi-phase optimization strategy (MOST) approach to optimize energy balance (EB) interventions in a sample of MD Anderson employees. (Pilot I) II. To explore the feasibility of using the MOST approach to optimize energy balance interventions in a sample of BRCA (BReast CAncer)-positive and Lynch syndrome positive individuals and their family members. (Pilot II) III. To explore the feasibility of using the MOST approach to optimize energy balance interventions in a sample of CLL (chronic lymphocytic leukemia) patients. (Pilot III)

SECONDARY OBJECTIVES:

I. To develop preliminary estimates of effect size and outcome variability for use in planning future studies. (Pilot I) II. To develop preliminary estimates of effect size and outcome variability for use in planning future studies. (Pilot II) III. To develop preliminary estimates of effect size and outcome variability for use in planning future studies. (Pilot III)

EXPLORATORY OBJECTIVES:

I. To examine relationship between individual-level (e.g., distress) and family-level (e.g., shared mutation status) variables that are specific to high-risk families and the effectiveness of energy balance interventions. (Pilot II)

OUTLINE: Participants are assigned to 1 condition in each component for a total of 16 groups using a randomized factorial design.

TELEPHONE COACHING VS EMAIL COACHING: Participants receive telephone coaching once per week for 16 weeks or 1 email per week for 16 weeks (with follow-up responses if the participant responds) from a coach trained in motivational interviewing.

TEXT MESSAGES: Participants receive daily text messages promoting adherence to diet and exercise recommendations daily 1-3 times per day or no text messages.

SOCIAL NETWORKING: Participants are invited to an online forum for study participants available for 16 weeks or do not receive an invitation for social networking.

SELF-MONITORING: Participants are asked to record their dietary intake 4-7 days per week or 1 day per week on a website or smartphone application (app).

After completion of study, patients are followed up at 4 months.

ELIGIBILITY:
Inclusion Criteria:

* PILOTS I, II AND III: Body mass index (BMI) of 25 or higher OR < 150 minutes of moderate to vigorous exercise per week OR < 5 servings of fruit and vegetables per day
* PILOTS I, II AND III: Capable of participating in moderate-vigorous unsupervised exercise
* PILOTS I, II AND III: Have a cellular telephone and are able and willing to send and receive text messages
* PILOTS I, II AND III: Able to read and write English
* PILOTS I, II AND III: Have access to internet
* PILOT II: BRCA positive OR Lynch syndrome positive individuals
* PILOT II (FAMILY MEMBER): Female and male biological and non-biological family members of BRCA-positive individuals OR Lynch syndrome positive individuals
* PILOT III: CLL survivors
* PILOT III: Has experienced fatigue within the past seven days

Exclusion Criteria:

* PILOTS I, II AND III: Unable to walk without crutches, walker, cane, or other assistive device
* PILOTS I, II AND III: Women who are pregnant (by self-report)
* PILOTS I, II AND III: Less than 3 months post-surgery
* PILOTS II and III: Currently receiving radiation therapy or cytotoxic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2014-09-17 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in waist circumference (Pilot I) | Baseline to 4 months post-intervention
  Expressed as the mean difference.
Change in waist circumference (Pilot II) | Baseline to 4 months post-intervention
  Expressed as the mean difference.

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Basen-Engquist, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Crane JC, Gordon MJ, Basen-Engquist K, Ferrajoli A, Markofski MM, Lee CY, Fares S, Simpson RJ, LaVoy EC. Relationships between T-lymphocytes and physical function in adults with chronic lymphocytic leukemia: Results from the HEALTH4CLL pilot study. Eur J Haematol. 2023 Jun;110(6):732-742. doi: 10.1111/ejh.13958. Epub 2023 Mar 31. PMID 36946440
- See also: M D Anderson Cancer Center — http://www.mdanderson.org